CLINICAL TRIAL: NCT03143855
Title: Phase I Drug Interaction and Subjective Effects of Compounds for Opioid Use Disorder
Brief Title: Drug Interaction and Subjective Effects of Compounds for Opioid Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20008062; U54DA038999 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Opioid Abuse; Opioid Dependence; Opioid-Related Disorders; Opioid Use
Keywords: oxycodone; lorcaserin; Belviq
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lorcaserin (Experimental)
  Interventions: Drug: Lorcaserin
- Control Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin will be administered at a dose of 10 mg twice daily for 5 days
  Arms: Lorcaserin
Drug: Placebo — Placebo will be administered twice daily for for 5 days
  Arms: Control Group

SUMMARY:
The overall goal of this project is to develop initial human data on effects of novel compounds on safety (interactions with oxycodone) and efficacy (subjective response to oxycodone) in non-treatment seeking opioid use disorder subjects. The compound to be studied will be the 5-HT2CR agonist lorcaserin. There are no known or reported adverse interactions between lorcaserin and oxycodone or other opioids.

DETAILED DESCRIPTION:
Lorcaserin is a serotonin (5-HT) 2C receptor agonist (Trade Name Belviq) approved for treatment of obesity. The study teams's preclinical research collaborators and others have shown that lorcaserin and other 5-HT2CR agonists have been shown to reduce drugs of abuse self-administration and cue reactivity in rodents including cocaine and nicotine. Recently, this data has been expanded to opioids. Rats trained to self-administer oxycodone showed a significant reduction in self-administration and oxycodone cue induced lever presses after lorcaserin administration.

This is a single center, double-blind, placebo-controlled, randomized, 1b/2a study. 18 subjects are planned. The following treatment regimens will be used:

Lorcaserin will be administered at a dose of 10mg twice daily. Placebo or Comparator - identical placebo capsules administered at the same time as lorcaserin.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, subjects must:

1. Males and females between 18 and 70 years-of-age.
2. Understand the study procedures and provide written informed consent.
3. Meet current DSM-5 criteria for opioid use disorder, at least moderate severity, but are not seeking treatment.
4. Have at least one positive urine drug screen for opioids during screening to document opioid use.
5. Have no clinically significant abnormalities in the judgment of the study physician in hematology and chemistry laboratory tests including liver function tests.
6. Have no contraindications for study participation as determined by medical history and physical examination.
7. Be able to demonstrate an understanding of study procedures and follow instructions including behavioral laboratory testing.
8. No pregnant or nursing women will be permitted in the study, and women must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device with spermicide, or condoms). Men will be advised to use condoms. All females must provide negative pregnancy urine tests before study entry, at each visit during the study, and at the end of study participation.

Exclusion Criteria:

In order to participate in the study, subjects must not:

1. Meet current DSM-5 diagnosis of any psychoactive substance use disorder other than opioids, marijuana, cocaine or nicotine. Diagnosis of mild to moderate use disorder for alcohol will not be considered exclusionary (SCID).
2. Have a current DSM-5 axis I psychiatric disorder other than substance use disorder including but not limited to Bipolar Disorder, Major Depressive Disorder, ADHD, or Schizophrenia or a neurological disorder requiring ongoing treatment and/or making study participation unsafe.
3. Have any previous medically adverse reaction to oxycodone or other opioids or lorcaserin.
4. Have any untreated clinically significant medical disorder including cardiovascular, pulmonary, CNS, hepatic, or renal disorder.
5. Have a history of seizures (excluding childhood febrile seizures), or loss of consciousness from traumatic injury for more than 30 minutes.
6. Have significant current suicidal or homicidal ideation or a history of suicide attempt within the past 6 months.
7. Have conditions of probation or parole requiring reports of drug use to officers of the court.
8. Have impending incarceration.
9. Have a positive HIV test by self-report or history.
10. Be pregnant or nursing or not using a reliable form of contraception if able to conceive. All females must provide negative pregnancy urine tests at screening, and daily after hospital admission.
11. Have any other illness, or condition, which in the opinion of the PI would preclude safe and/or successful completion of the study.
12. Have taken any investigational drug within 90 days prior to baseline.
13. Have an allergy to lorcaserin or oxycodone.
14. Have taken or are currently taking drugs that are know to inhibit cytochrome P450, CYP3A or CYP2D6.
15. ECG with QTc > 440ms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 participants signed the consent form however 5 participants were no shows for the initial visit at which ranndomization occurred.
Period: Overall Study
Arm/Group | Lorcaserin | Control Group
Started | 17 | 10
Completed | 12 | 6
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Participant experienced withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin | Control Group | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10.2) | 46 (8.8) | 48 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 11 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Response to Oxycodone Measured With 100 Millimeter Visual Analog Scale
Description: Drug liking is measured on a 100 millimeter visual analog rating with one end of the line representing a score of 0 for "not at all" and the other end being a score of 100 or extremely. Participants complete the rating 45 minutes after a 20 mg dose of oxycodone at baseline and after after 5 days of treatment.
Time Frame: Baseline to day 5
Population: Males and Females between ages 18 and 70 who meet criteria for opioid use disorder, at least moderate severity, but are not seeking treatment. Subjects diagnosed with a current psychiatric disorder or mental disorder including cardiovascular, pulmonary, CNS, hepatic or renal disorder are excluded from participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lorcaserin | Control Group
Number analyzed (Participants) | 11 | 6
units on a scale | -13.81 (31.7) | -9.67 (32.6)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Lorcaserin | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/12 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin (N=12) | Control Group (N=6)
Emesis (Psychiatric disorders) | 0 (0) | 1 (1) — Participant experienced withdrawal symptoms and receive Zofran. We felt it was not related to the study drug but was related to the participant taking more opioids than he told us which led to his withdrawal symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT03143855/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03143855/Prot_SAP_001.pdf